CLINICAL TRIAL: NCT05922982
Title: Norepinephrine Weaning Guided by the Hypotension Prediction Index in Vasoplegic Shock After Cardiac Surgery
Acronym: NORAHPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0046
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Vasoplegia; Shock; Norepinephrine; Surgery
Keywords: vasoplegia; shock; hypotension prediction index; Acumen; CABG; norepinephrine; surgery
MeSH Terms: conditions — Vasoplegia; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care arm (Active Comparator): MAP-based (MAP > 65 mmHg) norepinephrine weaning protocol
  Interventions: Drug: norepinephrine weaning protocol
- Experimental arm (HPI-guided) (Experimental): MAP-based (MAP > 65 mmHg) norepinephrine weaning protocol and guided by the HPI (HPI<80) delivered by the Acumen IQ medical device.
  Interventions: Drug: norepinephrine weaning protocol and guided by the HPI

INTERVENTIONS:
Drug: norepinephrine weaning protocol — MAP-based (MAP > 65 mmHg) norepinephrine weaning protocol
  Arms: Standard care arm
Drug: norepinephrine weaning protocol and guided by the HPI — MAP-based (MAP > 65 mmHg) norepinephrine weaning protocol and guided by the HPI (HPI<80) delivered by the Acumen IQ medical device.
  Arms: Experimental arm (HPI-guided)

SUMMARY:
In postoperative cardiac surgery under extracorporeal circulation, the patient may develop a vasoplegic syndrome, characterized by arterial hypotension (mean arterial pressure (MAP) < 65 mmHg); a decrease in vascular resistance and a cardiac output that may be normal or increased, and increased postoperative mortality/ International recommendations recommend the prescription of noradrenaline as a first-line treatment to reduce morbidity and mortality. However, excess norepinephrine or duration of exposure is also deleterious. The Acumen IQ device (Edwards Lifesciences) allows the calculation of a predictive index of arterial hypotension episodes (predictive hypotension index, HPI). HPI could improve norepinephrine weaning by preventing episodes of arterial hypotension or detecting preload dependence, thus avoiding the transient increase in norepinephrine during hypotension.

This is a single-center, prospective, open-label, randomized, controlled, 2-group, parallel, intention-to-treat study. The aim was to evaluate the superiority of a new decision algorithm, based on the HPI delivered by the Acumen IQ device, to reduce the duration of norepinephrine administration in post-cardiac surgery vasoplegic shock.

The duration of the interventional protocol is 72 hours. To evaluate the clinical impact of the protocol, the time of the study will be 30 days. Several follow-up visits will be performed (end-of-protocol day, discharge day, and at D30 of inclusion) to collect clinical, biological, and HPI monitoring data.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* The patient was hospitalized in the cardiothoracic-vascular and respiratory intensive care unit of Amiens-Picardy University Hospital.
* Patient scheduled for on-pomp cardiac surgery [coronary artery bypass grafting, valve replacement, ascending aorta replacement, or combined surgery (valve and bypass grafting)].
* Introduction of norepinephrine post-surgery for the treatment of vasoplegic syndrome.
* On-pomp cardiac surgery in less than 48 hours.
* Hemodynamically stable patient with MAP > 65 mmHg for more than 4 hours on noradrenaline
* Monitoring of MAP with a radial or femoral arterial catheter
* Social security beneficiary
* Signature of the consent to participate in the study by the patient, preoperatively

Exclusion Criteria:

* Permanent arrhythmia (atrial fibrillation, flutter, or frequent atrial extrasystoles).
* Treatment with dobutamine, epinephrine, or vasopressin analog
* Patients with preoperative chronic end-stage renal failure require postoperative extra-renal purification.
* Pregnant woman
* The patient is dependent on an internal or external pacemaker.
* Hypothermia < 36°.
* Patient under mechanical circulatory assistance after cardiac surgery.
* Hemorrhagic shock
* Patient under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the duration of norepinephrine administration between both groups | 72 hours
  The duration will be defined as the difference in time between the beginning of the study (day 0) and the end of the study protocol (day 3).

SECONDARY OUTCOMES:
Number of norepinephrine protocol weaning failures | 2 years
  Number of norepinephrine protocol weaning failures, defined as persistent norepinephrine delivery 72 hours after the start of inclusion
Prevalence of hypotensive episodes monitored by the Acumen IQ® device | 72 hours
  Hypotension is defined by the presence of a mean arterial pressure < 65 mmHg for a minimum duration of 30 seconds. Blood pressure must be invasive and monitored on the HemoSphere® monitor.
Frequency of hypotensive episodes monitored by the Acumen IQ® device | 72 hours
  Hypotension is defined by the presence of a mean arterial pressure < 65 mmHg for a minimum duration of 30 seconds. Blood pressure must be invasive and monitored on the HemoSphere® monitor.
Duration of hypotensive episodes monitored by the Acumen IQ® device | 72 hours
  Hypotension is defined by the presence of a mean arterial pressure < 65 mmHg for a minimum duration of 30 seconds. Blood pressure must be invasive and monitored on the HemoSphere® monitor.
NE total dose | 72 hours
  The NE (norepinephrine) total dose delivered during the research protocol phase (mg/kg) automatically calculated by the DianeRea® software (BowMedical, France).
Cumulative diuresis | 72 hours
  The Cumulative diuresis (ml.kg.h) during protocol completion (H0 to H72) or when norepinephrine weaning is considered successful.
Volume of administrated fluids | 72 hours
  Cumulative volume of administration of crystalloids, colloids, or blood products during protocol or when NE weaning is considered as successful.
Total dose of vasoactive drugs | 72 hours
  Vaso-active drugs. The total dose of vasoactive drug initiation or reintroduction of NE after the weaning protocol calculated by the NEE and the VIS.
Number of stroke | 72 hours
  Stroke (Any embolic, thrombotic or haemorrhagic cerebral event with persistent residual motor, sensory or cognitive dysfunction (eg, hemiplegia, hemiparesis, aphasia, sensory deficit, impaired memory) diagnosed on a cerebral scanner)
Number of myocardial infarction | 72 hours
  Myocardial infarction diagnosed by the clinical presentation, serial changes on 12-lead electrocardiographic suggesting infarction, and rise in cardiac markers (preferably cardiac troponins) with at least one value above the 99th percentile of the upper reference limit.
Number of resuscitated cardiac arrest | 72 hours
  Cessation of mechanical cardiac activity confirmed by the absence of clinical signs of blood flow
Number of acute kidney injury | 72 hours
  Increase in serum creatinine of over 27 μmol/L within 48 hours or diuresis lower than 0.5 mL/kg/hour (KDIGO Guidelines).
Number of mesenteric ischaemia | 72 hours
  Mesenteric ischaemia confirmed by imaging or exploratory laparotomy and/or ischaemic colitis confirmed by gastrointestinal endoscopy or exploratory laparotomy
Number of in-hospital mortality. | 72 hours
  Mortality from surgery to hospital discharge
Number of 30 days hospital mortality | 30 days
  Mortality after surgery until 30 days follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyls C, Lefebvre T, Mollet N, Boussault A, Meynier J, Abou-Arab O, Mahjoub Y. Norepinephrine weaning guided by the Hypotension Prediction Index in vasoplegic shock after cardiac surgery: protocol for a single-centre, open-label randomised controlled trial - the NORAHPI study. BMJ Open. 2024 Jun 26;14(6):e084499. doi: 10.1136/bmjopen-2024-084499. PMID 38926148